CLINICAL TRIAL: NCT00637819
Title: A Randomized, Double-Blind, Placebo Controlled Clinical Trial of Leflunomide in Systemic Lupus Erythematosus (SLE)
Brief Title: Leflunomide in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Iris Chan/Study Director, sanofi-aventis
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HWA486_6014
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Systemic Lupus Eythematosus (SLE)
MeSH Terms: interventions — Leflunomide

INTERVENTIONS:
Drug: Leflunomide — A loading dose of LEF 100mg daily for 3 days, followed by LEF 20mg daily for the remainder of the study or matching placebo
  Other Names: Arava

SUMMARY:
A pilot study to evaluate the efficacy and safety of leflunomide in SLE patients with active disease who are refractory to cyclophosphamide

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the revised ACR criteria for SLE with either evidence of active disease according to SLE Disease Activity Index (SLEDAI)

Exclusion Criteria:

* Patients who are pregnant or nursing women, or those with life threatening disease
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-01; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
number of patients who are able to achieve complete remission, defined as a SLEDAI of 0 | 52 weeks

SECONDARY OUTCOMES:
number of patients who are able to achieve partial remission, as defined by a SLEDAI of 1-3 | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iris Chan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Hong Kong, Hong Kong